CLINICAL TRIAL: NCT00999752
Title: A 25 Week, Open Label Study to Determine the Effects of Nebivolol When Added to Hydrochlorothiazide on Diastolic Function and Arterial Stiffness in African Americans With Hypertension
Brief Title: Study to Determine the Effects of Nebivolol and Hydrochlorothiazide in African Americans With Hypertension
Acronym: NASAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InVasc Therapeutics, Inc. (Industry)
Responsible Party: Bobby V. Khan, MD PhD, InVasc Therapeutics, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AVR-2009-02 (BYS-MD-27)
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: Hypertension; African Americans; Arterial Stiffness; Vascular Resistance
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Nebivolol to reach blood pressure control
  Interventions: Drug: Nebivolol
- Arm B (Active Comparator): Hydrochlorothiazide for blood pressure control
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Nebivolol — 5mg/day with increase to 10 mg/day to reach blood pressure <140/90
  Other Names: Bystolic
  Arms: Arm A
Drug: Hydrochlorothiazide — Hydrochlorothiazide 25 mg/day
  Other Names: HCTZ
  Arms: Arm B

SUMMARY:
The main purpose of this study is to evaluate the effects of Nebivolol and Hydrochlorothiazide on blood pressure in African Americans with high blood pressure.

DETAILED DESCRIPTION:
Many blood pressure medications are not effective in African American men and women. The two lower chambers of the heart contract to pump blood to the body. The lower chambers have to relax so they can refill with blood to pump out again. Many patients with high blood pressure have stiffness in the lower chambers which prevents the heart from relaxing so it can properly fill with blood. Some patients with the stiffness in the lower chambers of the heart will develop heart failure.

The study is to test whether or not Nebivolol (Bystolic)and a diuretic Hydrochlorothiazide (HCTZ) will help the heart relax so the heart can properly fill and prevent stiffness of the lower heart chambers.

ELIGIBILITY:
Inclusion Criteria:

* Known Hypertension by history
* Self-described African American

Exclusion Criteria:

* Uncontrolled Diabetes Mellitus (HbA1C>10)
* Known CAD, Cerebrovascular Disease, PVD or Renovascular Disease
* Liver disease
* Chronic Renal Disease
* Uncontrolled Hypertension (>199 systolic and/or >115)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Changes in systolic and diastolic blood pressure after treatment with nebivolol and reaching normal blood pressure <140/90 | Every visit for 25 weeks (9 study visits)

SECONDARY OUTCOMES:
Differences after nebivolol treatment on diastolic function as measured by tissue doppler imaging (ECHO), arterial compliance and stiffness and vascular nitric oxide availability determined by neutrophil function | At the begining and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bobby V Khan, MD PhD, Principal Investigator — InVasc Therapeutics, Inc.
Locations (1):
- Atlanta Vascular Research Foundation, Tucker, Georgia, United States